CLINICAL TRIAL: NCT01656018
Title: Phase 1 Open Label Safety, Acceptability, Pharmacokinetic and ex Vivo Pharmacodynamic Study of TMC278 Long Acting (LA) Administered Intramuscularly to HIV-1 Seronegative Individuals
Brief Title: A Study to Evaluate Safety, Acceptability, Pharmacokinetics, and ex Vivo Pharmacodynamics of TMC278 Long Acting Formulation in HIV-1 Seronegative Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR100803; TMC278-MWRI-01 (Other: Janssen Research and Development, LLC)
Record Dates: First submitted 2012-07-31; First posted 2012-08-02 (Estimated); Last update posted 2016-04-07 (Estimated); Status verified 2016-04

CONDITIONS: Healthy
Keywords: Healthy; TMC278; Human Immunodeficiency Virus Type 1; HIV-1; Pharmacokinetics; Ex-vivo pharmacodynamics
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Rilpivirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (10):
- Arm 1A (Experimental): Female participants will receive a single dose of long acting TMC278 1200 mg intramuscularly (IM) at baseline (Day 0) in Arm 1A.
  Interventions: Drug: TMC278, Long acting (LA)
- Arm 1B (Experimental): Male participants will receive a single dose of long acting TMC278 1200 mg IM at baseline in Arm 1B.
  Interventions: Drug: TMC278, Long acting (LA)
- Arm 2A (Experimental): Female participants will receive a single dose of long acting TMC278 600 mg IM at baseline in Arm 2A.
  Interventions: Drug: TMC278, Long acting (LA)
- Arm 2B (Experimental): Male participants will receive a single dose of long acting TMC278 600 mg IM at baseline in Arm 2B.
  Interventions: Drug: TMC278, Long acting (LA)
- Arm 3A (Experimental): Female participants will receive 3 bi-monthly injections of long acting TMC278 1200 mg IM at baseline, Months 2 and 4 in Arm 3A.
  Interventions: Drug: TMC278, Long acting (LA)
- Arm 3B (Experimental): Male participants will receive 3 bi-monthly injections of long acting TMC278 1200 mg IM at baseline, Months 2 and 4 in Arm 3B.
  Interventions: Drug: TMC278, Long acting (LA)
- Arm 4A (Experimental): Female participants will receive a single dose of long acting TMC278 1200 mg IM at baseline followed by TMC278 900 mg at Months 2 and 4 in Arm 4A.
  Interventions: Drug: TMC278, Long acting (LA)
- Arm 4B (Experimental): Male participants will receive a single dose of long acting TMC278 1200 mg IM at baseline followed by TMC278 900 mg at Months 2 and 4 in Arm 4B.
  Interventions: Drug: TMC278, Long acting (LA)
- Arm 5A (Experimental): Female participants will receive a single dose of long acting TMC278 1200 mg IM at baseline followed by TMC278 600 mg at Months 2 and 4 in Arm 5A.
  Interventions: Drug: TMC278, Long acting (LA)
- Arm 5B (Experimental): Male participants will receive a single dose of long acting TMC278 1200 mg IM at baseline followed by TMC278 600 mg at Months 2 and 4 in Arm 5B.
  Interventions: Drug: TMC278, Long acting (LA)

INTERVENTIONS:
Drug: TMC278, Long acting (LA) — TMC278 long acting will be administered IM to the participants as follows: a single dose of TMC278 600 mg will be administered at baseline in Arm 2A and Arm 2B; at Months 2 and 4 in Arm 5A and Arm 5B. A single dose of TMC278 900 mg will be administered at Months 2 and 4 in Arm 4A and Arm 4B. A single dose of TMC278 1200 mg will be administered at baseline in Arm 1A, Arm 1B; Arm 3A, Arm 3B, Arm 4A, Arm 4B, Arm 5A and Arm 5B; at Months 2 and 4 in Arm 3A and Arm 3B.
  Other Names: TMC278

SUMMARY:
The purpose of this study is to evaluate the safety, acceptability, pharmacokinetics (what the body does to the medication), and ex vivo (tested outside the body) pharmacodynamics (what the medication does to the body) of TMC278 long acting (slowly effective after initial dosage and maintaining its effects over a long period of time) when administered as an intramuscular (ie, in to the muscle) injection in adult participants who are seronegative for human immunodeficiency virus type 1 (HIV-1).

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), multi-arm (more than one treatment group), dose-ranging study (clinical study where different doses of study medication are tested against each other) to evaluate the safety, acceptability, pharmacokinetics, and ex vivo pharmacodynamics of a single and multiple intramuscular injections of long acting TMC278 to human immunodeficiency virus type 1 (HIV-1) seronegative (having a negative serum reaction) male and female participants. The study consists of 3 phases including screening phase, treatment phase, and the follow up phase (approximately 4 to 6 months after the first dose of study medication). In treatment phase, enrolled participants will be divided in to 2 arms, ie, Arm A (female participants) which will be further divided in to Arm 1A, Arm 2A, Arm 3A, Arm 4A, and Arm 5A with 12 female participants per arm; and Arm B (male participants) which will be further divided in to Arm 1B, Arm 2B, Arm 3B, Arm 4B, and Arm 5B with 6 male participants per arm. Safety evaluations will include assessment of adverse events, clinical laboratory tests, electrocardiogram, physical examination, and vital signs which will be monitored throughout the study. The total duration of study for each participant will be approximately 5 to 7 months.

ELIGIBILITY:
Inclusion Criteria:

* Human immunodeficiency virus type 1 (HIV-1) seronegative at screening and enrollment
* Not pregnant or breastfeeding females
* Agrees to protocol-defined method of contraception
* Abstinence from insertion of anything in rectum (eg, medication, enema, penis, or sex toy) for 72 hours before and 72 hours after each rectal biopsy visit
* Abstinence from insertion of anything in vagina (eg, tampon, medication, douche, penis, or sex toy) for 72 hours before and 72 hours after each cervical and vaginal biopsy visit

Exclusion Criteria:

* Post-exposure prophylaxis for HIV exposure within 6 months prior to screening and known HIV-infected partners
* Use of systemic immunomodulatory medications within the 4 weeks prior to the enrollment
* Use of vaginally or rectally administered medications or products (including condoms) containing Nonoxynol-9 (N-9) within the 4 weeks prior to the enrollment
* Abnormalities of the cervical, vaginal, or colorectal mucosa, or significant symptom(s), which in the opinion of the clinician represents a contraindication to protocol-required biopsies
* History of recurrent urticaria
* History of or electrocardiogram demonstrating prolonged QT interval
* History of significant gastrointestinal bleeding

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2012-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | Up to 280 days
Number of participants who would consider using long acting TMC278 for Human immunodeficiency virus (HIV) prevention in the future | Up to 280 days

SECONDARY OUTCOMES:
TMC278 concentration in plasma | Up to 280 days
TMC278 concentration in endocervical fluid | Up to 280 days
TMC278 concentration in vaginal fluid | Up to 280 days
TMC278 concentration in rectal fluid | Up to 280 days
TMC278 concentration in cervical tissue | Up to 280 days
TMC278 concentration in vaginal tissue | Up to 280 days
TMC278 concentration in rectal tissue | Up to 280 days

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research and Development, LLC Clinical Trial, Study Director — Janssen Research and Development LLC
Locations (1):
- Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Derived] McGowan I, Dezzutti CS, Siegel A, Engstrom J, Nikiforov A, Duffill K, Shetler C, Richardson-Harman N, Abebe K, Back D, Else L, Egan D, Khoo S, Egan JE, Stall R, Williams PE, Rehman KK, Adler A, Brand RM, Chen B, Achilles S, Cranston RD. Long-acting rilpivirine as potential pre-exposure prophylaxis for HIV-1 prevention (the MWRI-01 study): an open-label, phase 1, compartmental, pharmacokinetic and pharmacodynamic assessment. Lancet HIV. 2016 Dec;3(12):e569-e578. doi: 10.1016/S2352-3018(16)30113-8. Epub 2016 Sep 16. PMID 27658864